CLINICAL TRIAL: NCT02664025
Title: The Benefits of Simulation in Teaching Vaginal Examination for Women During Labor: a Randomized Controlled Study
Brief Title: Simulation in Teaching Vaginal Examination
Acronym: VE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: VE
Record Dates: First submitted 2016-01-22; First posted 2016-01-26 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Healthy
Keywords: teaching vaginal examination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- simulation group (Active Comparator): Interns will carry out 10 VE on a simulator
  Interventions: Procedure: vaginal examination simulator
- Control group (No Intervention): Interns who will not perform any simulated VE

INTERVENTIONS:
Procedure: vaginal examination simulator
  Arms: simulation group

SUMMARY:
Teaching technical skills during medical training can lead to some issues, which can concern ethical or medico-legal risks. In this context, the vaginal examination (VE) is specific because it concerns the genital area and it interferes with obstetrical management.

ELIGIBILITY:
Inclusion Criteria:

* Interns who finished their study in faculty of medicine
* Interns who never performed VE before
* Interns who accept to participate in the study

Exclusion Criteria:

* Interns who refuse to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-03; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
the improvement of vaginal examination accuracy score after practical training on simulators | 5 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes